CLINICAL TRIAL: NCT03457571
Title: Clinical Observational Study: IBD Patients With Restless-legs-syndrome and Iron Deficiency Syndrome
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Janek Becker, MD, Charite University, Berlin, Germany
Other Study IDs: EA4/132/13
Record Dates: First submitted 2018-03-01; First posted 2018-03-07 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Inflammatory Bowel Diseases; Restless Legs Syndrome; Iron-deficiency
MeSH Terms: conditions — Inflammatory Bowel Diseases; Restless Legs Syndrome; Anemia, Iron-Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with inflammatory bowel disease, such as Crohn´s disease or ulcerative colitis, have recurring episodes of abdominal pain, diarrhea and loss of weight. Besides this other clinical symptoms are possible e.g. deficiency syndromes such as iron deficiency. Iron deficiency usually attended by symptoms like hair loss, pale skin, loss of concentration or fatigue. In some cases iron deficiency can lead to neurological manifestations such as restless-legs-syndrome (RLS). Restless legs syndrome is a neurological disorders which is accompanied by substantial urge to move legs or other parts of the body and unpleasant sensations.

Aim of this study is to to investigate the prevalence of RLS in patients with inflammatory bowel disease and furthermore evaluate the effect of iron supplementation in patients with iron deficiency and concomitant RLS.

DETAILED DESCRIPTION:
Restless legs syndrome (RLS) is a common neurological disease significantly impacting live quality. Two recent studies from North America and Japan revealed a surprisingly high prevalence for RLS in Crohn´s disease and ulcerative colitis (30% and 21%, respectively). The underlying cause for this high prevalence remains elusive at this point.

To address this gap, a cohort of 353 IBD patients from a tertiary IBD centre was prospectively evaluated by our IBD team as well as by the colleagues from neurology. IBD patients (age ≥ 18 years) presenting at our IBD outpatient clinic (tertiary referral center) between February 2014 and February 2015 were prospectively recruited for the study after written consent. The study was approved (16 January 2014) by the ethics committee of the Charité - Universitätsmedizin Berlin, Campus Benjamin Franklin (reference EA4/132/13). Patients were screened for symptoms of iron deficiency (ID) and RLS by a self-developed questionnaire and explored for RLS symptoms by a gastroenterologist. When at least one symptom of RLS was present, patients were referred to a neurologist for RLS or differential diagnosis.

Additionally patients with RLS symptoms were screened for iron-, folic acid- and vitamin B12-deficiency. If a deficiency was detected, patients were substituted. In patients with deficiencies, follow-up visits were scheduled at week 4 and 11 after starting supplementation. Follow-up visits were conducted by the neurologist and the IRLS was performed in all patients at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Written consent
* Age > 18
* Inflammatory bowel disease

Exclusion Criteria:

* <18 years
* No written consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with inflammatory bowel disease in IBD outpatient clinic (tertiary referral center) in Germany
Sampling Method: Probability Sample
Enrollment: 353 (Actual)
Dates: Start 2014-02-01 (Actual); Primary Completion 2015-02-28 (Actual); Study Completion 2015-04-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of RLS in IBD | 1 year

SECONDARY OUTCOMES:
Prevalence of clinically relevant RLS in IBD | 1 year

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Becker J, Berger F, Schindlbeck KA, Poddubnyy D, Koch PM, Preiss JC, Siegmund B, Marzinzik F, Maul J. Restless legs syndrome is a relevant comorbidity in patients with inflammatory bowel disease. Int J Colorectal Dis. 2018 Jul;33(7):955-962. doi: 10.1007/s00384-018-3032-8. Epub 2018 Apr 3. PMID 29610943